CLINICAL TRIAL: NCT02475642
Title: Pulmonary Vein Isolation With Versus Without Continued Antiarrhythmic Drug Treatment in Subjects With Recurrent Atrial Fibrillation: A Prospective 2-Centre Randomized Controlled Clinical Study (POWDER-AF)
Brief Title: Pulmonary Vein Isolation With Versus Without Continued Antiarrhythmic Drug Treatment in Subjects With Recurrent Atrial Fibrillation
Acronym: POWDER-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VZW Cardiovascular Research Center Aalst (Other)
Collaborators: AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POWDER-AF01
Record Dates: First submitted 2015-06-03; First posted 2015-06-19 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI-ADT (Active Comparator): discontinue antiarrhythmic drugs at 3 months post PVI
  Interventions: Other: PVI-ADT
- PVI+ADT (Active Comparator): discontinue antiarrhythmic drugs at 12 months post PVI
  Interventions: Other: PVI+ADT

INTERVENTIONS:
Other: PVI-ADT — Discontinue antiarrhythmic drugs at randomisation (3 months post ablation). As per the eligibility criteria, all patients randomised are taking either Flecainide, Cibenzoline, Propafenon, Sotalol or Amiodarone. These are discontinued at the moment of randomisation in this arm
  Arms: PVI-ADT
Other: PVI+ADT — Discontinue antiarrhythmic drugs 9 months after randomisation (12 months post ablation). As per the eligibility criteria, all patients randomised are taking either Flecainide, Cibenzoline, Propafenon, Sotalol or Amiodarone. These are continued in this arm until 9 months post randomisation at which point they are stopped
  Arms: PVI+ADT

SUMMARY:
The purpose of this study is to compare the efficacy and safety of PV isolation with continued antiarrhythmic drug treatment (PVI+ADT) to PV isolation without continued ADT (PVI-ADT) in patients undergoing treatment for symptomatic recurrent AF.

DETAILED DESCRIPTION:
Subjects that underwent PV isolation for paroxysmal or non-longstanding persistent AF and are free of arrhythmia at the end of the 3-month blanking period while taking ADT. Eligible subjects who sign the study informed consent form will be randomized into one of two study arms:

PVI+ADT Group: continue ADT through 9 months follow-up PVI-ADT Group: no ADT through 9 months follow up

ELIGIBILITY:
Inclusion Criteria:

* patient has continued (IC or III) ADT throughout the 3-month blanking
* patient is free of symptomatic and asymptomatic AF (as evidenced by 1-day Holter) at the 3-month visit
* drug-resistant (at least one class IC or III) symptomatic AF was the primary indication for prior PV isolation
* in the three months prior to PVI, at least one episode of symptomatic or asymptomatic AF
* PV isolation was performed according to the standards set forward by the Task Force Document (sedation or general anesthesia)
* PV isolation was the only target for ablation (except for cavotricuspid (CTI) ablation if documented AFL)
* PV isolation was performed by point-by-point irrigated radio frequency (RF) guided by contact-force (Biosense) (10-30gr-continuous lesion)
* PV isolation (i.e. entry block) was verified in each vein after a waiting time and adenosine (with continued RF if acute reconnection)
* Signed Patient Informed Consent Form.
* Age 18 years or older.
* Able and willing to comply with all follow-up testing and requirements.

Exclusion Criteria:

* Longstanding persistent atrial fibrillation (>12 months of continuous AF)
* Previous ablation for AF
* left atrium (LA) size > 55 mm
* left ventricular ejection fraction (LVEF) < 40%
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* coronary artery bypass graft (CABG) procedure within the last six months
* Awaiting cardiac transplantation or other cardiac surgery
* Documented left atrial thrombus on imaging
* Diagnosed atrial myxoma
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable) or breastfeeding
* Acute illness or active systemic infection or sepsis
* Unstable angina
* Uncontrolled heart failure
* Myocardial infarction within the previous two (2) months
* History of blood clotting or bleeding abnormalities
* Contraindication to anticoagulation therapy (ie, heparin or warfarin)
* Life expectancy less than 12 months
* Enrollment in any other study evaluating another device or drug
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction
* Patients not taking any class IC or III ADT at 3 months after PV isolation
* No documentation of entry block at initial PV isolation - no waiting time or adenosine.
* Additional linear ablation or defractionation during the initial procedure (except for CTI ablation for documented or induced cavo-tricuspid isthmus dependent flutter).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by freedom of arrhythmia recurrence | 9 months
  Arrhythmia recurrence rate at 1 year post ablation (9 months post randomization)
Safety as measured by drug discontinuation | 9 months
  Number of participants with any adverse events at 1 year post ablation (9 months post randomization) leading to drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, MD, PhD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (2):
- Belgium (2):
  - OLV Hospital, Aalst
  - AZ St Jan, Bruges